CLINICAL TRIAL: NCT06012110
Title: Transcutaneous Electrical Stimulation for Spasticity in Patients With Primary Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-219-NSU
Record Dates: First submitted 2023-08-14; First posted 2023-08-25 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Primary Lateral Sclerosis
MeSH Terms: conditions — Motor Neuron Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcutaneous electrical stimulation to reduce spasticity in PLS (Experimental): Primary lateral sclerosis (PLS) is a progressive upper motor neuron neurodegenerative disorder. A hallmark of PLS is a presentation with lower extremity stiffness and spasticity as well as bulbar involvement. The investigators will be performing a preliminary study designed to assess transcutaneous electrical stimulation (tES), a non-pharmacological and non-invasive modality used in spinal cord injury and multiple sclerosis patients, as a treatment for reducing spasticity in the lower extremities and increasing mobility in patients with PLS.
  Interventions: Device: Transcutaneous electrical stimulation

INTERVENTIONS:
Device: Transcutaneous electrical stimulation — While participants are supine with a pillow placed below the knees for comfort, one 30-minute transcutaneous electrical stimulation session will be performed at a frequency of 50 Hz, pulse width of 400 microseconds and individualized amplitude will be completed.

SUMMARY:
The goal of this clinical trial is to determine if non-invasive electrical stimulation, using an electric stimulator placed on the skin of the patients back and abdomen for 30 minutes can reduce muscle spasms (spasticity) and improve walking function in patients with primary lateral sclerosis. Participants will attend one in-person clinic visit and participate in one telephone interview 24 hours after the treatment. The clinic visit will include pre-intervention, treatment and post-intervention assessments. The assessments will consist of a complete physical exam by the clinic neurologist followed by assessments and scoring of spasticity, deep tendon reflexes, gait quality, gait speed, gait endurance and balance. Patient's will rate their perceived spasticity pre, immediately post and 24 hours post treatment.

The treatment involves one 30-minute electrical stimulation session, which includes application of electrode pads to the patients back and abdomen. The patient will lay supine (on their back) with a pillow placed under their knees for comfort. The pads will then be connected to an FDA approved electrical stimulator. The electrical stimulator will be turned on and current adjusted to the individual patient based on small muscle contractions in their legs. Once the current is set, the patient will lay supine for 30 minutes. After 30 minutes, the device will be turned off and electrode pads removed.

DETAILED DESCRIPTION:
Objective: The primary aim of this preliminary pilot study is to assess the clinical effects of transcutaneous electrical stimulation (tES) in reducing spasticity in the lower extremities and increasing mobility in patients with Primary Lateral Sclerosis (PLS).

Study population: 6 patients with a confirmed diagnosis of PLS aged 18-90

Design:

Each enrolled participant will attend one in-person clinic visit and participate in one telephone interview 24 hours post-treatment.

The clinic visit will include pre-intervention, treatment and post-intervention assessments. The assessments will consist of a complete physical exam by the clinic neurologist followed by assessments and scoring of spasticity, deep tendon reflexes, gait quality, gait speed, gait endurance and balance. The patients will rate their perceived spasticity pre, immediately post and 24 hours post treatment.

Treatment will include a 30-minute transcutaneous electrical stimulation (tES) session where tES will be applied through two sets of electrodes positioned adjacent to the T11/T12 spinous processes and a second pair of electrodes placed para-umbilically on the lower abdomen. A current-controlled electrical stimulator will be used to deliver charge-balanced symmetrical, biphasic rectangular pulses to the paraspinal electrodes as the anode for the first phase and as the cathode for the second phase of the stimulation phase.

Electrode placement will be verified by applying electrical stimulation to elicit mild posterior root-muscle (PRM) contractions in the L2-S2 innervated rectus femoris, biceps femoris, tibialis anterior, and triceps surae muscle group bilaterally with the participants relaxed in the supine position. This will be determined by palpation at the patellar and achilles tendons of both sides. While the participants remain supine, the stimulator will be set to continuous mode to deliver stimulation at a frequency of 50 Hz and pulse width of 400 microseconds, then the stimulation amplitude will be slowly increased from 0 milliamp (mA) to an amplitude that may generate minor paraesthesias (slight tingling sensations) in some individuals in the bilateral L2-S2 lower extremity dermatomes but below the level that elicited posterior motor root (PMR) contraction responses. The stimulation amplitude will be individually assessed and set for each participant, and the stimulation amplitude upper limit will be no more than 90% of the lowest PRM response for each participant. After this 30-minute tES session, the tES unit will be turned off, the electrodes removed, and the participants assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary lateral sclerosis by the treating neurologist
* Ambulatory with or without a assistive device or orthotic

Exclusion Criteria:

* History of cancer in the lumbar or thoracic spine
* History of surgery with hardware in the lumbar or thoracic spine
* Acute lower back pathology
* Current pregnancy
* History of implantable cardiac device
* Diagnosis of significant cognitive impairment by the treating physician
* History of seizures or diagnosis of epilepsy
* Open wound at location of electrodes
* Complete loss of sensation at the area of electrode placement

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale | through study completion, an average of 1 year
  6 category ordinal scale (minimum value = 0 maximum value = 4) that measures spasticity where higher scores indicate greater spasticity

SECONDARY OUTCOMES:
Deep Tendon Reflex Scale | through study completion, an average of 1 year
  5 point ordinal scale recorded as a number from 0-4 where 2 is normal and any number above or below this is abnormal.
10-meter walk test (10MWT) | through study completion, an average of 1 year
  The 10MWT measures gait speed where the time it takes patient to cover a distance of 6 meters is recorded in m/s.
6 minute walk test (6MWT) | through study completion, an average of 1 year
  The 6MWT assesses overall gait function and endurance. The total distance travelled in 6 minutes is recorded in feet.
Tinetti Performance Oriented Mobility Assessment | through study completion, an average of 1 year
  3 point ordinal scale that ranges from 0-2 with a total possible score of 28 that measures gait quality and balance. Higher scores indicate improved gait and balance.
0-10 numeric rating scale | through study completion, an average of 1 year
  Patients will self rate their spasticity on a scale of 0-10 with 0 = no spasticity and 10 = worst possible spasticity.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Locatelli, MD, MPH, Principal Investigator — Nova Southeastern University; Alan Boruch, DO, PhD, Principal Investigator — Northeast Regional Medical Center / A.T. Still University
Locations (1):
- NSU Health Neuroscience Institute, Davie, Florida, United States

IPD SHARING:
Plan to Share IPD: No
This study will provide pilot data to establish a larger, more robust study. The data will be kept internally.

REFERENCES:
- [Background] Feldman EL, Goutman SA, Petri S, Mazzini L, Savelieff MG, Shaw PJ, Sobue G. Amyotrophic lateral sclerosis. Lancet. 2022 Oct 15;400(10360):1363-1380. doi: 10.1016/S0140-6736(22)01272-7. Epub 2022 Sep 15. PMID 36116464
- [Background] Nashold BS Jr, Friedman H. Dorsal column stimulation for control of pain. Preliminary report on 30 patients. J Neurosurg. 1972 May;36(5):590-7. doi: 10.3171/jns.1972.36.5.0590. No abstract available. PMID 5026545
- [Background] Cook AW, Weinstein SP. Chronic dorsal column stimulation in multiple sclerosis. Preliminary report. N Y State J Med. 1973 Dec 15;73(24):2868-72. No abstract available. PMID 4543587
- [Background] Lin A, Shaaya E, Calvert JS, Parker SR, Borton DA, Fridley JS. A Review of Functional Restoration From Spinal Cord Stimulation in Patients With Spinal Cord Injury. Neurospine. 2022 Sep;19(3):703-734. doi: 10.14245/ns.2244652.326. Epub 2022 Sep 30. PMID 36203296
- [Background] Hofstoetter US, Freundl B, Danner SM, Krenn MJ, Mayr W, Binder H, Minassian K. Transcutaneous Spinal Cord Stimulation Induces Temporary Attenuation of Spasticity in Individuals with Spinal Cord Injury. J Neurotrauma. 2020 Feb 1;37(3):481-493. doi: 10.1089/neu.2019.6588. Epub 2019 Aug 9. PMID 31333064
- [Background] Hofstoetter US, Freundl B, Lackner P, Binder H. Transcutaneous Spinal Cord Stimulation Enhances Walking Performance and Reduces Spasticity in Individuals with Multiple Sclerosis. Brain Sci. 2021 Apr 8;11(4):472. doi: 10.3390/brainsci11040472. PMID 33917893
- [Background] Turner MR, Barohn RJ, Corcia P, Fink JK, Harms MB, Kiernan MC, Ravits J, Silani V, Simmons Z, Statland J, van den Berg LH; Delegates of the 2nd International PLS Conference; Mitsumoto H. Primary lateral sclerosis: consensus diagnostic criteria. J Neurol Neurosurg Psychiatry. 2020 Apr;91(4):373-377. doi: 10.1136/jnnp-2019-322541. Epub 2020 Feb 6. PMID 32029539
- See also: Link to electrical stimulator utilized in this study — https://compasshealthbrands.com/products?pSearch=intensity%20select%20combo%20II